CLINICAL TRIAL: NCT03795610
Title: Phase 2 Window of Opportunity Study of IPI-549 in Patients With Locally Advanced HPV+ and HPV- Head and Neck Squamous Cell Carcinoma
Brief Title: IPI-549 in Patients With Locally Advanced HPV+ and HPV- Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assuntina G. Sacco, MD (Other)
Collaborators: The V Foundation for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, Assuntina G. Sacco, MD, Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 172058
Record Dates: First submitted 2018-12-21; First posted 2019-01-08 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer; Head and Neck Carcinoma; Head and Neck Cancer Stage IV; Head and Neck Cancer Stage III; HPV-Related Carcinoma; HPV-Related Malignancy; HPV-Related Squamous Cell Carcinoma
Keywords: HPV positive; HPV negative; HPV-; HPV+; PI3K-γ; microenvironment; immunotherapy; tumor; resection; PI3K; cancer; carcinoma; malignancy; head; neck; throat; esophageal; nasopharyngeal; nasopharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Neoplasms; Carcinoma | interventions — IPI-549

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm A: IPI-549 40 mg PO qdaily (Experimental): Patients enrolled in Arm A will receive IPI-549 40 mg by mouth daily for at least 14 days
  Interventions: Drug: IPI-549

INTERVENTIONS:
Drug: IPI-549 — 40mg by mouth (PO) every day (QD) for at least 14 days
  Other Names: Eganelisib

SUMMARY:
The purpose of this study is to investigate how effective the study drug IPI-549 is against types of cancers. IPI-549 is considered experimental because it is not approved by the US Food and Drug Administration (FDA) for the treatment of cancer.

Patients will be treated with 2 weeks of IPI-549, a specific PI3Kγ inhibitor. Tumor tissue for research purposes through core biopsies will be obtained prior to initiation of IPI-549 and at surgery.

DETAILED DESCRIPTION:
This is a phase 2 window of opportunity trial in patients with locally advanced head and neck cancer. A key objective is to provide the first proof that macrophage phenotype switching can be accomplished in humans and lay the groundwork for future trials of this novel approach to immune therapy. Patients who are candidates for surgical resection will be enrolled and treated with 2 weeks of IPI-549, a specific PI3Kγ inhibitor. Tumor tissue for research purposes through core biopsies will be obtained prior to initiation of IPI-549 and at surgery.

The study team hypothesizes that mRNA signatures of immune response will be increased in IPI-549-treated patients. For the efficacy endpoints, RECISTv1.1 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Have locally advanced that is amenable to surgical resection
* Must be able to swallow tablets
* Must be able to undergo a core tumor biopsy.
* Must have adequate organ function.

Exclusion Criteria:

* Diagnosis of cutaneous squamous cell carcinoma (SCC) or Epstein-Barr virus (EBV) related nasopharynx cancer.
* Planned major surgery within 4 weeks prior to initiation of study drug
* Patients treated with chemotherapy, biologic therapy, or other investigational agent within < 28 days of starting study drug
* History of infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C virus (HCV)
* On going treatment with chronic immunosuppressants (e.g., cyclosporine) or systemic steroids
* Prior surgery or gastrointestinal dysfunction that may affect drug absorption (e.g. gastric bypass surgery, gastrectomy)
* Female subjects who are pregnant or breastfeeding
* Concurrent active malignancy other than nonmelanoma skin cancer, carcinoma in situ of the cervix, or prostate intraepithelial neoplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

REFERENCES:
- [Background] Kaneda MM, Cappello P, Nguyen AV, Ralainirina N, Hardamon CR, Foubert P, Schmid MC, Sun P, Mose E, Bouvet M, Lowy AM, Valasek MA, Sasik R, Novelli F, Hirsch E, Varner JA. Macrophage PI3Kgamma Drives Pancreatic Ductal Adenocarcinoma Progression. Cancer Discov. 2016 Aug;6(8):870-85. doi: 10.1158/2159-8290.CD-15-1346. Epub 2016 May 13. PMID 27179037
- [Background] Kaneda MM, Messer KS, Ralainirina N, Li H, Leem CJ, Gorjestani S, Woo G, Nguyen AV, Figueiredo CC, Foubert P, Schmid MC, Pink M, Winkler DG, Rausch M, Palombella VJ, Kutok J, McGovern K, Frazer KA, Wu X, Karin M, Sasik R, Cohen EE, Varner JA. PI3Kgamma is a molecular switch that controls immune suppression. Nature. 2016 Nov 17;539(7629):437-442. doi: 10.1038/nature19834. Epub 2016 Sep 19. PMID 27642729
- [Background] De Palma M, Lewis CE. Macrophage regulation of tumor responses to anticancer therapies. Cancer Cell. 2013 Mar 18;23(3):277-86. doi: 10.1016/j.ccr.2013.02.013. PMID 23518347
- [Background] Gabrilovich DI, Ostrand-Rosenberg S, Bronte V. Coordinated regulation of myeloid cells by tumours. Nat Rev Immunol. 2012 Mar 22;12(4):253-68. doi: 10.1038/nri3175. PMID 22437938
- [Background] Schmid MC, Avraamides CJ, Dippold HC, Franco I, Foubert P, Ellies LG, Acevedo LM, Manglicmot JR, Song X, Wrasidlo W, Blair SL, Ginsberg MH, Cheresh DA, Hirsch E, Field SJ, Varner JA. Receptor tyrosine kinases and TLR/IL1Rs unexpectedly activate myeloid cell PI3kgamma, a single convergent point promoting tumor inflammation and progression. Cancer Cell. 2011 Jun 14;19(6):715-27. doi: 10.1016/j.ccr.2011.04.016. PMID 21665146
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: IPI-549 40 mg PO Qdaily
Started | 16
Completed | 10
Not Completed | 6
Not completed — Screen Failure (Did not meet inclusion/exclusion) | 4
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure (Unknown) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm A: IPI-549 40 mg PO Qdaily
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 1
  Unknown or Not Reported | 2
Cancer Type [Count of Participants; unit: Participants]
  Nasal cavity | 1
  Oral cavity | 4
  Oropharynx | 5

OUTCOME MEASURES:

1. Primary Outcome: Participants Experiencing Adverse Events
Description: To determine safety and tolerability of IPI-549 in patients with locally advanced HNSCC.
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: IPI-549 40 mg PO Qdaily
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | Arm A: IPI-549 40 mg PO Qdaily
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: IPI-549 40 mg PO Qdaily (N=10)
Sepsis (Infections and infestations) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: IPI-549 40 mg PO Qdaily (N=10)
Gastrointestinal disorders (Gastrointestinal disorders) | 8 (14)
General disorders and administration site conditions (General disorders) | 4 (4)
Immune system disorders (Immune system disorders) | 1 (1)
Investigations (Investigations) | 1 (2)
Nervous system disorders (Nervous system disorders) | 3 (5)
Psychiatric disorders (Psychiatric disorders) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Vascular disorders (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT03795610/Prot_SAP_002.pdf
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT03795610/ICF_001.pdf